CLINICAL TRIAL: NCT03857633
Title: The Process of Inflammation in the Development of Myocardial Fibrosis in Chronic Kidney Disease and End Stage Renal Failure - A Longitudinal Cohort Study Assessing Myocardial Fibrosis Development Using Cardiac MRI Correlated With Monocyte and Biochemical Profile Analysis During Transition to Renal Replacement Therapy
Brief Title: MRI Assessment of Myocardial Fibrosis Associated With Monocyte Phenotype in End Stage Renal Failure
Acronym: CM3
Status: Withdrawn | Type: Observational
Why Stopped: Suspended
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18HH4615; 221424 (Other: IRAS ID)
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Myocardial Fibrosis; End Stage Renal Failure on Dialysis; Chronic Kidney Disease, Stage IV (Severe); Chronic Kidney Disease Stage V; Heart Failure
Keywords: Cardiac MRI; Myocardial Fibrosis; End Stage Renal Failure; Monocyte Subsets; Renal Replacement Therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood and Serum Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre Dialysis (CKD Stage 4/5): Patients recruited from low clearance clinic with advanced CKD (stage 4/5). Patients will undergo Cardiac MRI 1 - With Gadolinium Contrast at the time of recruitment and Cardiac MRI 2 - With Gadolinium Contrast at time of commencement on renal replacement therapy. Patients will have Peripheral Whole Blood Samples taken at defined intervals.
  Interventions: Diagnostic Test: Cardiac MRI 1 - With Gadolinium Contrast; Diagnostic Test: Cardiac MRI 2 - With Gadolinium Contrast; Diagnostic Test: Peripheral Whole Blood Samples
- Haemodialysis Dialysis (CDK Stage 5d): Patients started on Haemodialysis will have Cardiac MRI 3 - With Gadolinium Contrast after 6 months of therapy. Patients will have Peripheral Whole Blood Samples taken at defined intervals.
  Interventions: Diagnostic Test: Cardiac MRI 3 - With Gadolinium Contrast; Diagnostic Test: Peripheral Whole Blood Samples
- Peritoneal Dialysis (CDK Stage 5d): Patients started on Peritoneal Dialysis will have Cardiac MRI 3 - Without Gadolinium Contrast after 6 months of therapy. Patients will have Peripheral Whole Blood Samples taken at defined intervals.
  Interventions: Diagnostic Test: Cardiac MRI 3 - Without Gadolinium Contrast; Diagnostic Test: Peripheral Whole Blood Samples

INTERVENTIONS:
Diagnostic Test: Cardiac MRI 1 - With Gadolinium Contrast — Cines for cardiac function and volumes, T2 myomaps, Resting perfusion and strain analysis, Tagging (strain), T1 myomaps, Late gadolinium enhancement
  During the MRI scan participants would be required perform a short period of low intensity exercise involving peddling on an adapted cycle for 10-15 minutes to provide additional data on cardiac function under exertion.
  Groups: Pre Dialysis (CKD Stage 4/5)
Diagnostic Test: Cardiac MRI 2 - With Gadolinium Contrast — Cines for cardiac function and volumes, T2 myomaps, Resting perfusion and strain analysis, Tagging (strain), T1 myomaps, Late gadolinium enhancement
  During the MRI scan participants would be required perform a short period of low intensity exercise involving peddling on an adapted cycle for 10-15 minutes to provide additional data on cardiac function under exertion.
  Groups: Pre Dialysis (CKD Stage 4/5)
Diagnostic Test: Cardiac MRI 3 - Without Gadolinium Contrast — Cines for cardiac function and volumes, T2 myomaps, Resting perfusion and strain analysis, Tagging (strain), T1 myomaps.
  During the MRI scan participants would be required perform a short period of low intensity exercise involving peddling on an adapted cycle for 10-15 minutes to provide additional data on cardiac function under exertion.
  Groups: Peritoneal Dialysis (CDK Stage 5d)
Diagnostic Test: Cardiac MRI 3 - With Gadolinium Contrast — Cines for cardiac function and volumes, T2 myomaps, Resting perfusion and strain analysis, Tagging (strain), T1 myomaps, Late gadolinium enhancement
  During the MRI scan participants would be required perform a short period of low intensity exercise involving peddling on an adapted cycle for 10-15 minutes to provide additional data on cardiac function under exertion.
  Groups: Haemodialysis Dialysis (CDK Stage 5d)
Diagnostic Test: Peripheral Whole Blood Samples — 20ml EDTA whole blood samples - collected sequentially during study - max 8 time points

SUMMARY:
Firstly, this study aims to understand how cardiac fibrosis mediated by inflammatory microvascular disease evolves during advanced chronic kidney disease and end stage renal failure and importantly how this changes with commencement on renal replacement therapy (haemodialysis and peritoneal dialysis) using sequential cardiac MRI imaging. This method of imaging is non-invasive, provides significantly more data than echocardiography, is reproducible and accurate, has been validated in numerous studies and does not involve exposure to ionising radiation.

Secondly, this study aims to examine the changes in monocyte subsets and biochemical profile in peripheral blood prior to, during and after commencement on renal replacement therapy.

The investigators hypothesis would be that renal failure causes alteration in monocyte subset phenotype resulting in increased circulating inflammatory monocytes (human CD14high CD16high), initiating pro-inflammatory cytokine expression and thereby accelerating inflammatory cardiovascular disease and development of myocardial fibrosis.

DETAILED DESCRIPTION:
There is significant excess of cardiac mortality in patients with end stage renal failure (ESRF) - 15 to 20% relative increased risk of cardiac death compared to the normal population. 20-30% of patients on renal replacement therapy (RRT) die from a cardiac cause (UK Renal Registry Data, 2016). However, only 30% have macrovascular disease at the time of autopsy. There is therefore a significant component of cardiac morbidity and mortality in this population that is mediated by microvascular disease and cardiac fibrosis. This includes abnormal myocardial remodelling, increased ventricular stiffness and ventricular hypertrophy, with development of arrhythmia and cardiac failure as well as increased atherosclerotic disease burden. Renal replacement therapy in itself also induces a pro-inflammatory response in patients increasing cardiac risk and there is poor understanding as to how to mediate this risk.

There is a lack of evidence in how to manage both patients and the RRT process to minimise the risk of patients developing cardiac disease. The mechanisms underlying this enhanced risk are not fully understood nor explained by traditional cardiovascular risk factors. The investigators propose to study the mechanism by which this might be mediated.

The investigators have previously reported alterations in monocyte subset populations in CKD patients that importantly predict CVD events. Furthermore, the investigators have shown that dyslipidaemia influences monocyte/macrophage phenotypes. The investigators propose an important interaction exists between chronic inflammation in the uraemic state, dyslipidaemia and the formation of deleterious monocyte/macrophage phenotypes that accelerates atherosclerosis. Cardiac MRI has been used in recent years to accurately assess the degree of cardiac fibrosis in end stage renal failure.

This clinical study builds on previous clinical and non-clinical studies at Imperial College London by unifying basic science, animal models and imaging studies into the clinical context of end stage renal failure. Increased understanding of the changes in cardiac function related to development of end stage renal failure and commencement on renal replacement therapy will provide significant and novel opportunities to optimise the management of patients in the pre-dialysis setting and prevent cardiovascular complications caused by long term renal replacement therapy.

This clinical observational study will involve the recruitment of 30 participants from general nephrology services at Imperial College Healthcare NHS Trust at CKD stage 4/5 with progressive decline in renal function (anticipated start on renal replacement therapy within 6 months). Participants will be divided into two cohorts of haemodialysis and peritoneal dialysis to enable comparison between the renal replacement modalities. As part of participants recruitment they will undergo comprehensive medical assessment and will remain under the follow-up of the renal team at frequent intervals.

Enrolled participants will undergo cardiac MRI imaging at three time points - First when initially recruited at CKD4/5, second at the point of commencement on renal replacement therapy (~6 months) and third after a further 6 months on renal replacement therapy. MRI results will be analysed at these time points for development of fibrotic and function change.

In partnership with MRI imaging patients will have blood samples collected at the same time intervals for analysis of blood count, biochemical markers, monocyte and lipid phenotypes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of Chronic Kidney Disease stage 4 and above
2. Patients with a progressive decline in renal function with a expectation to require future renal replacement therapy or currently on renal replacement therapy (Haemodialysis or Peritoneal Dialysis)
3. Exclusion of macrovascular cardiac disease within the last 3 years
4. Access for haemodialysis planned via tunnelled central venous catheter

Exclusion Criteria:

1. Age under eighteen
2. Patients with a diagnosis of Diabetes Mellitus
3. Untreated macrovascular cardiac disease or Acute Coronary syndrome within 6 months of recruitment
4. Previous or current treatment with immunosuppressive/modulatory therapy
5. Current Malignancy
6. Current use of Metformin
7. Pregnancy
8. Contraindication to MRI Imaging
9. Patients lacking capacity or unable to consent and non-English language speakers
10. Immediate modality switch after commencement on renal replacement therapy i.e. transplantation
11. Plan for treatment centre change/move outside of Imperial College Healthcare NHS Trust following commencement on renal replacement therapy
12. Patients currently participating in an active CTIMP trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced and progressive Chronic Kidney Disease (Stage 4/5) - under low clearance follow-up who are expected to start renal replacement therapy (either haemodialysis or peritoneal dialysis) within 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
The development and modulation of myocardial fibrosis and change in cardiac function with CKD progression and commencement on renal replacement therapy | 18 Months
  Cardiac MRI assessment of the evolution of myocardial fibrosis and cardiac function using sequential contrast enhanced CMR imaging (at three time points) during transition to end stage renal failure and commencement on renal replacement therapy

SECONDARY OUTCOMES:
Change in monocyte subsets and biochemical profile in peripheral blood with CKD progression and commencement on renal replacement therapy | 18 Months
  Assessment of change in monocyte subset (phenotype and function), plasma cytokine levels and lipid profile in sequential blood samples collected during transition from advanced CKD to commencement on renal replacement therapy correlated with myocardial fibrosis and cardiovascular risk.

CONTACTS AND LOCATIONS:
Overall Officials: Neill Duncan, MBBS FRCP, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No